CLINICAL TRIAL: NCT06967701
Title: Informatics-Based Digital Intervention to Promote Safe Exercise in Middle-Aged Adults With Type 1 Diabetes and Other Absolute Insulin Deficiency Diabetes - A Pilot Efficacy Study
Brief Title: Building and Sustaining Exercise Habits for Adults With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Garrett I Ash, PhD, Assistant Professor of Medicine, Biomedical Informatics, and Data Science, Yale University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000039977; K01DK129441 (NIH)
Record Dates: First submitted 2025-05-03; First posted 2025-05-13 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes (T1D); Latent Autoimmune Diabetes in Adult (LADA); Pancreatitis
Keywords: exercise; physical activity; mobile phone; health coaching; fitness watch
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Pancreatitis; Motor Activity | interventions — Resistance Training; Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Monitoring (Active Comparator): Wear a fitness watch and keep daily health diary
  Interventions: Behavioral: Self-monitoring
- Exercise program (Experimental): Participants will receive a free Garmin smartwatch and a free program membership providing exercise coaching + personalized feedback about the relationship among their insulin, carbohydrates, exercise, sleep, and blood sugar.
  Interventions: Behavioral: Exercise program

INTERVENTIONS:
Behavioral: Exercise program — Participants will receive a free Garmin smartwatch and a free program membership providing exercise coaching + personalized feedback about the relationship among their insulin, carbohydrates, exercise, sleep, and blood sugar.
  Arms: Exercise program
Behavioral: Self-monitoring — Wear a fitness watch and keep daily health diary
  Arms: Self-Monitoring

SUMMARY:
The challenges of living with type 1 diabetes often stand in the way of getting enough exercise. Continuous blood sugar monitoring has revolutionized type 1 diabetes care but remains underutilized to sustainably support exercise and related behaviors. This remote participation-based research will develop a mobile application that delivers personalized encouragement and data-driven health insights based upon patterns in blood sugar, exercise, mood, and sleep, to assist people with type 1 diabetes in exercising more frequently and confidently. You do not need to live in Connecticut to participate, as there will be no required in-person visits during the study.

ELIGIBILITY:
Inclusion criteria:

* 30-65 years old inclusive
* Diagnosis with type 1 diabetes (T1D) or other insulin deficiency diabetes (latent autoimmune disease of adulthood, diabetes secondary to pancreatitis)
* Less than 1.0 exercise sessions per week
* Smartphone ownership
* English literacy
* Under regular care by a healthcare provider (1+ appointments per year)
* Home Broadband wireless Internet or cell phone network
* Using continuous glucose monitor (CGM) and sharing data with medical record for at least 6 weeks
* Using insulin pump or pen and sharing data with medical record for at least 6 weeks

Exclusion criteria:

* Diabetic ketoacidosis not clearly related to pump site failure in past 6 months
* >1 episode of severe hypoglycemia (altered mental and/or physical status requiring assistance from another person for recovery) in past 6 months
* A1c ≥10.0%
* Resting blood pressure >160mmHg systolic or >100 mmHg diastolic.
* Myocardial infarction or angina in past 12 months
* Uncontrolled arrhythmia (e.g., atrial fibrillation with rapid ventricular response, new onset atrial fibrillation, ventricular tachycardia, escape rhythms)
* Congestive heart failure (stage 3 or 4)
* Exercise-induced asthma (not controlled on inhalers)
* Chronic obstructive pulmonary disease (requiring home oxygen)
* Renal failure
* Pregnancy
* Cognitive impairment
* Severe retinopathy or neuropathy.
* Other chronic disease or physical disability that would influence exercise intervention (e.g., recent spinal surgery)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Weekly exercise duration | 20 weeks
  Minutes/week. Measured by blinded hip watch and periodic interviews. 0 minutes/week is the lowest value, 150 minutes/week meets clinically recommended amounts.

SECONDARY OUTCOMES:
Weekly exercise volume | 20 weeks
  Kilocalories, determined by minutes and intensity. Measured by blinded hip watch and periodic interviews. A person achieving 150 minutes per week will achieve around 1,200 - 2,000 kilocalories per week.
Weekly exercise days | 20 weeks
  Days/week. Measured by blinded hip watch and periodic interviews. 0 days/week is the lowest value, 3-7 days/week meets clinically recommended amounts.
Glucose | 20 weeks
  The measurable range is 20-400 mg/dL. It is quantified by average levels, time above/within/below the target range of 70-180 mg/dL, and coefficient of variation.
Body mass index | 20 weeks
  Calculated from body weight and height (kilograms per meters squared)
Waist circumference | 20 weeks
  Measured in centimeters at umbilicus
Blood pressure | 20 weeks
  Systolic and diastolic values in mmHg. Values above 130 / 85 are considered hypertensive range. Measured on home monitor in duplicate
Sleep disturbance | 20 weeks
  NIH PROMIS (Patient-Reported Outcomes Measurement Information System) sleep disturbance survey. Scores given in t-score reflecting value relative to population.
Sleep-related impairment | 20 weeks
  NIH PROMIS (Patient-Reported Outcomes Measurement Information System) sleep-related impairment survey. Scores given in t-score reflecting value relative to population.
Affective motivation states | 20 weeks
  Cravings for Rest and Volitional Energy Expenditure (CRAVE) survey of motivation states for physical activity. Scores range from 0 (not at all) to 10 (more than ever).
Fear of hypoglycemia | 20 weeks
  Survey with subscales of fear-related behavior and worry respectively. Scores range from 0 (never) to 4 (almost always).
Fear of hyperglycemia | 20 weeks
  Survey with subscales of glucose decisions, lifestyle decisions, and worry. Scores range from 1 (never) to 5 (always).
Exercise self-efficacy | 20 weeks
  Asks about confidence to achieve exercise goals. Scores range from 0 (not confident) to 10 (very confident).
Exercise self-regulation | 20 weeks
  Survey of reasons for motivation to exercise. Participants rate possible reasons with scores ranging from 1 (not at all true) to 7 (very true).

CONTACTS AND LOCATIONS:
Overall Officials: Garrett Ash, PhD, CSCS, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes